CLINICAL TRIAL: NCT03331640
Title: A Health Service Research Study to Investigate Survival of Metastatic Pancreatic Cancer Patients After Sequential Chemotherapy: An AIO Phase II Cross Over Trial (PANTHEON)
Brief Title: A Health Service Research Study to Investigate Survival of Metastatic Pancreatic Cancer Patients After Sequential Chemotherapy
Acronym: PANTHEON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AIO-PAK-0116
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — IFL protocol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFF (Experimental)
  Interventions: Drug: OFF
- FOLFIRI (Experimental)
  Interventions: Drug: FOLFIRI Protocol

INTERVENTIONS:
Drug: OFF — OFF:
  5-FU 2000 mg/m2 as 24 hour infusion + Na folinic acid 200 mg/m2 on D1, 8, 15, 22 Oxaliplatin 85 mg/m2 on D8, 22 3 weeks rest after D22; Cycle q42d
  Arms: OFF
Drug: FOLFIRI Protocol — Irinotecan 180 mg /m2 5-FU 400 mg/m2 (bolus) + 2400 mg/m2 as 46 hour infusion Na folinic acid 200 mg/m2 Cycle q2w
  Arms: FOLFIRI

SUMMARY:
The aim of the study is to assess the efficacy of second and third line therapies (OFF vs. FOLFIRI) in a sequential cross-over design in patients pretreated with nab-paclitaxel/gemcitabine first line.

DETAILED DESCRIPTION:
Secondary objectives are assessment of safety and feasibility of the sequential cross-over treatment approach for advanced treatment lines in PDAC. 204 patients will be randomized into the treatments arms. Cross-over will take place after progress during second line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry
3. Unresectable adenocarcinoma of the pancreas previously treated in the palliative setting with gemcitabine and nabpaclitaxel (Abraxane®)
4. Adequately documented recurrence and disease status after/under 1st line (Best response, duration of treatment, time to progression, preexisting PNP and other side effects)
5. Radiologically confirmed disease progression during 1st-line therapy and measurable reference cancer site(s) as defined by RECIST1.1
6. Randomization and start of 2nd-line treatment possible within 4 weeks after radiologically documented disease progression during 1st-line therapy
7. ECOG performance status 0-2
8. No prior radiotherapy
9. Adequate blood count, liver-enzymes, and renal function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * AST (SGOT)/ALT (SGPT) < 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be < 5x ULN
   * Serum creatinine CL ≥ 60 mL/min calculations according to local standard
   * Bilirubin < 3 ULN
10. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥ 60 years old and no menses for ≥ 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry
11. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Serious cardiovascular disease (eg, unstable coronary artery disease or myocardial infarction within 3 months prior to study start)
2. Preexisting polyneuropathy (PNP) ≥ grade 3 [National Cancer Institute Common Toxicity Criteria grade 3 or 4 sensory or motor neuropathy]
3. Prior or concurrent malignancy (other than pancreatic cancer) which either progresses or requires active treatment. Exceptions are: basal cell cancer of the skin
4. History of DPD deficiency
5. Morbus Gilbert
6. History of hypersensitivity to any of the study drugs or any of the constituents of the products
7. Medication that is known to interfere with any of the agents applied in the trial
8. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year)
9. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
10. Any medical condition that contraindicates dosing with any of the IMPs or constitutes a safety risk for the patient including but not limited to:

    1. chronic inflammatory bowel disease and/or bowel obstruction.
    2. active uncontrolled infection
    3. clinically significant bleeding or bleeding diathesis
    4. clinically significant stomatitis
    5. active ulceration of the gastrointestinal tract
11. Previous enrollment or randomization in the present study (does not include screening failure)
12. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG
13. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Progression-free survival during 2nd line therapy (PFS2) | 49 months
  Progression-free survival time from randomization till progress during second line therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Praxis für Innere Medizin, Friedrichshafen, Germany

REFERENCES:
- See also: Homepage of the AIO (Arbeitsgemeinschaft Internistische Onkologie in der Deutschen Krebsgesellschaft e.V.) — http://www.aio-portal.de